CLINICAL TRIAL: NCT06522386
Title: GATE1: A Multicenter Phase II Study of Pirtobrutinib, Rituximab and Venetoclax Combination Therapy for Patients With Previously Untreated Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry); Genentech, Inc. (Industry); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0220; NCI-2024-06175 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — pirtobrutinib; Rituximab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pirtobrutinib, Rituximab and Venetoclax combination (Experimental)
  Interventions: Drug: Pirtobrutinib; Drug: Rituximab; Drug: Venetoclax

INTERVENTIONS:
Drug: Pirtobrutinib — Given by mouth
Drug: Rituximab — Given by vein (IV)
  Other Names: Rituxan
Drug: Venetoclax — Given by mouth
  Other Names: ABT-199; GDC-0199

SUMMARY:
Primary Objectives:

To estimate the percent of participants who achieve a best response of complete response by the end of the PRV combination therapy in the induction therapy phase in patients with previously untreated MCL.

DETAILED DESCRIPTION:
Secondary Objectives:

* To evaluate the objective response rate to PRV combination therapy in patients with previously untreated MCL.
* To evaluate the duration of response in patients with an objective response to PRV combination therapy.
* To evaluate the progression-free survival and overall survival in patients treated with PRV combination therapy.
* To evaluate the safety profile of PRV combination therapy in patients with previously untreated MCL.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Confirmed pathology diagnosis of MCL with t(11;14)(q13;q32) translocation and/or cyclin D1 overexpression (e.g., positive immunohistochemistry staining).
3. MCL cells are CD20 positive (e.g., positive staining on immunohistochemistry or flow cytometry).
4. No prior MCL-directed systemic treatment (such as chemotherapy, immunotherapy, targeted therapy, and cellular therapy) or radiotherapy.

   NOTE: A short course of corticosteroids (e.g., ≤ 1 week of intravenous or ≤ 2 weeks of oral) given for acute MCL-related symptoms or impending severe organ dysfunction is allowed, but a washout period of 3 days is required before registration.
5. Have a clinical indication to treat (e.g., B symptoms, or symptomatic or progressive lymphadenopathy or hepatosplenomegaly, or cytopenia caused by MCL, etc.).
6. ECOG performance status (PS) 0-2 (Appendix I).
7. Evaluable disease, i.e., ANY of the following:

   * Measurable lymph node or extranodal lesion with at least one dimeson > 1.5 cm
   * Spleen size > 15 cm if spleen is involved by MCL (based on imaging or biopsy)
   * WBC > 15,000/µL if peripheral blood is involved by MCL (based on flow cytometry)
   * Bone marrow involvement by MCL (> 10% of cellularity)
   * Endoscopically visible lesion that is biopsy-proven to be involved by MCL
8. Meet ALL following criteria in lab values obtained ≤ 14 days prior to registration:

   * Absolute neutrophil count (ANC) ≥ 1000/µL without growth factor support
   * Platelet count ≥ 75,000/µL without transfusion support (≥ 50,000/µL if there is evidence of bone marrow involvement by MCL or splenomegaly due to MCL)
   * Hemoglobin ≥ 8.0 g/dL without transfusion support
   * Prothrombin (PT) or international normalized ratio (INR) ≤ 1.5 × upper normal limit (ULN)
   * Activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) ≤ 1.5 × ULN
   * Total bilirubin ≤ 1.5 × ULN, or ≤ 3 × ULN if there is evidence of parenchymal liver involvement by MCL; patients with Gilbert's syndrome or hemolysis are eligible if direct bilirubin is ≤ 1.5 × ULN
   * Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 3 × ULN, or ≤ 5 × ULN if there is evidence of parenchymal liver involvement by MCL
   * Creatinine clearance > 50 mL/min using the Cockcroft-Gault formula (Appendix II)
9. Left ventricular ejection fraction by ECHO or MUGA ≥ 50% (must be within 12 months prior to registration).
10. Able to understand and voluntarily sign an IRB-approved informed consent form.
11. Willing to provide mandatory research blood, bone marrow, lymphoma biopsy tissue, and saliva specimens for correlative research.
12. Willing to return to enrolling institution for follow-up.
13. Negative serum pregnancy test done ≤ 7 days prior to registration, for persons of childbearing potential, defined as post menarche and not postmenopausal (i.e., ≥ 2 years of non-therapy-induced amenorrhea) or surgically sterile (e.g., post-hysterectomy, bilateral salpingectomy, or oophorectomy).
14. Persons of reproductive potential and their partners must agree to use highly effective birth control methods for the duration of study treatment and for 1 month (30 days) following the last dose of pirtobrutinib and/or venetoclax and for 12 months following the last dose of rituximab (Appendix III).
15. Males must agree to not donate sperms for the duration of study treatment and for 3 months following the last dose of any study drug.

Exclusion Criteria:

1. CNS involvement by MCL (e.g., any parenchymal, leptomeningeal, CSF, cranial nerve, or spinal cord or nerve root involvement).
2. Pregnant or plan to become pregnant during study treatment or within 1 month following the last dose of pirtobrutinib and/or venetoclax or within 12 months following the last dose of rituximab; or breast-feeding or plan to breastfeed during study treatment or within 1 week following the last dose of pirtobrutinib and/or venetoclax or within 6 months following the last dose of rituximab.
3. Malabsorption syndrome or other condition that precludes enteral route of administration.
4. Any of the following medication requirement or recent use:

   * Use of a strong or moderate cytochrome P450 (CYP) 3A inhibitor or inducer ≤ 7 days prior to registration
   * Anticipated requirement of a strong CYP3A inhibitor or inducer during the study that cannot be substituted
   * Use of grapefruit or grapefruit products, Seville oranges or products from Seville oranges, or star fruit ≤ 3 days prior to registration, or planned use during the study
   * Anticipated requirement of a strong P-gp inhibitor during the study
   * Anticoagulation with a vitamin K antagonist ≤ 7 days prior to registration or anticipated use during the study
5. Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
6. History of a bleeding disorder (e.g., hemophilia, von Willebrand disease, etc.) or active bleeding.
7. Active or recent infections, including but not limited to:

   * Active infections requiring treatment (such as systemic antibiotics, antivirals, or antifungals) ≤ 7 days prior to registration
   * History of a positive COVID-19 (SARS-CoV-2) test (nucleic acid or antigen) within 4 weeks prior to registration, or presence of continued COVID-19-related clinically relevant symptoms or COVID-19-related significant pulmonary infiltrates in patients with a history of COVID-19 disease
   * Human Immunodeficiency Virus (HIV) positive NOTE: Patients who have tested positive for Human Immunodeficiency Virus (HIV) are excluded due to potential drug-drug interactions between anti-retroviral medications and pirtobrutinib and risk of opportunistic infections with both HIV and irreversible BTK inhibitors. For patients with unknown HIV status, HIV testing will be performed at Screening and result should be negative for the patient to be eligible.
   * Known active Cytomegalovirus (CMV) infection
   * Hepatitis B virus (HBV): Patients with positive hepatitis B surface antigen (HBsAg) are excluded. Patients with positive hepatitis B core antibody (anti-HBc) and negative HBsAg require HBV polymerase chain reaction (PCR) evaluation. Patients who are HBV PCR positive will be excluded. Due to rituximab's black box warning for Hepatitis B reactivation, patients with positive hepatitis B core antibody (anti-HBc) should have prophylactic therapy with an approved nucleos(t)ide analogue to prevent reactivation.
   * Hepatitis C virus (HCV): If hepatitis C antibody result is positive, patient will need to have a negative result for hepatitis C ribonucleic acid (RNA). Patients who are hepatitis C RNA positive will be excluded.
8. Uncontrolled cardiovascular disease including but not limited to:

   Uncontrolled hypertension (SBP > 160 mmHg or DBP > 110 mmHg despite of 3 different classes of full dose anti-hypertensives medications) History of myocardial infarction ≤ 3 months prior to registration Unstable angina or acute coronary syndrome ≤ 2 months prior to registration New York Heart Association (NYHA) Class III or IV or symptomatic congestive heart failure or dilated cardiomyopathy Uncontrolled or symptomatic arrhythmias NOTE: Patients with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker
9. Prolongation of QT interval corrected for heart rate (QTcF, calculated using Fridericia's Formula: QTcF=QT/∛RR) > 470 msec.

   NOTE: Correction for widened QRS complex (e.g., with pacing, or underlying bundle branch block, etc) allowed (e.g., "Adjusted QTcF" = measured QTcF - [measured QRS - 90 ms]). Correction of suspected drug induced QTcF prolongation can be attempted at the investigator's discretion and only if clinically safe to do so with either discontinuation of the offending drug or switch to another drug not known to be associated with QTcF prolongation.
10. History of cerebral vascular accident ≤ 6 months prior to registration.
11. Oxygen dependent lung disease (such as interstitial lung disease or COPD).
12. Ongoing inflammatory bowel disease (such as ulcerative colitis) requiring active treatment.
13. Psychiatric illness/social situations that would limit compliance with study requirements.
14. Major surgery ≤ 28 days prior to registration.
15. Vaccination with a live vaccine ≤ 28 days prior to registration.
16. Another primary malignancy (other than localized non-melanotic skin cancer or carcinoma in situ of the cervix or breast) that is not in remission or requires ongoing treatment (except for adjuvant hormonal therapy for adequately treated nonmetastatic breast or prostate cancer), or limits expected survival to ≤ 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wang, MD, MS, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org